## **The Effects of Dance for Breast Cancer Patients Undergoing Surgical Treatment**

**ID:** 74502023.7.0000.5432

## The Effects of Dance for Breast Cancer Patients Undergoing Surgical Treatment

Introduction: Breast cancer treatment can lead to changes in self-image, emotional and functional loss. Physiotherapy in the postoperative period of oncological surgeries has the main objectives of avoiding complications such as adherent scars which can compromise the range of movement of a limb involved, optimize function, promote function, promote muscle strength gain, maintain proper body posture, reduce skin and fascia adherence, and optimize the aesthetic result. Despite the patients are highly informed about the importance of physical activity, demotivation is a major barrier to continuing treatment. Dance is one of the activities that has been gaining ground and has the main benefit of rehabilitation of lost or impaired movements after surgery, in a playful way, through supervised and specialized follow-up for each patient. There are few randomized studies on the effects of dance on breast cancer patients undergoing surgical treatment. patients undergoing surgical treatment. The hypothesis is that dance will will improve range of motion, strength, functionality, quality of life, reduce pain and fatigue for breast cancer patients undergoing surgical treatment. Objectives: To evaluate the effects of dance as a therapeutic resource for breast cancer patients undergoing surgical treatment on: shoulder range of motion, overall muscle strength, fatigue, respiratory muscle strength, functionality, pain and quality of life. Method: This is a non-randomized randomized clinical trial, with pre- and post-intervention evaluation and prospective data collection. The following will be used for pre-intervention assessment: goniometry, dynamometry, manovacuometry, 6-minute walk test, fatigue and quality of life questionnaire, as well as a pain assessment scale. After 16 weeks, the same variables will be assessed.